CLINICAL TRIAL: NCT05683769
Title: Can microRNA Help to Differentiate Erosive Hand Osteoarthritis From Psoriatic Arthritis?
Brief Title: microRNA in Erosive Hand Osteoarthritis and Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: University of Siena (Other)
Responsible Party: Principal Investigator, fioravanti antonella, Principal Investigator, University of Siena
Other Study IDs: miRNA EHOA vs PsA
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Erosive Osteoarthritis; Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- erosive hand osteoarthritis: EHOA was diagnosed according to the American College of Rheumatology (ACR) criteria and to the presence of the classical central erosion in at least two IP joints. Further inclusion criteria were the availability of plain radiography of both hands performed in the previous 6 months. Plain radiographs of both hands were collected and scored by two readers according to Kallman's classification in a blind observation.
  Interventions: Genetic: miRNA
- psoriatic arthritis: PsA was diagnosed following the CASPAR classification guidelines and only patients with the peripheral arthritis pattern were considered; all PsA group had also the diagnosis of psoriasis confirmed by an expert dermatologist. These patients had also to be naive to conventional and biologic disease-modifying anti-rheumatic drugs (DMARDs) or have withdrawn any DMARDs for at least three months, because of inadequate response or intolerance.
  Interventions: Genetic: miRNA
- Control Group: The control group was represented by healthy volunteers age-and sex-matched to study patients and were recruited among the hospital staff; HC did not exhibit symptoms or signs attributable to OA, psoriasis, as well as to autoimmune disorders and systemic inflammatory arthropathies.
  Interventions: Genetic: miRNA

INTERVENTIONS:
Genetic: miRNA — Assessment of miRNA, as potential biomarkers to discriminate erosive hand osteoarthritis from psoriatic arthritis

SUMMARY:
Erosive osteoarthritis of the hand (EHOA) is a rare subset of HOA that affects mainly postmenopausal middle-aged women, featured by prominent signs of inflammation, severe progression, and typical radiographic changes of the interphalangeal (IP). It is presently debated whether EHOA is an advanced stage of the classical HOA or a separate entity with peculiar inflammatory features, which can mimic chronic arthritis such as psoriatic arthritis (PsA). PsA is a chronic immune-mediated inflammatory arthropathy, that affects 14.0-22.7% of patients with psoriasis. It is a highly heterogeneous disease, whose clinical features often vary from peripheral arthritis, to spinal spondylitis, and/or asymmetrical synovitis, enthesitis, dactylitis. As no gold-standard diagnostic test for PsA exists, the diagnosis is based on different patterns of clinical, radiological and serological markers included in the classification criteria for psoriatic arthritis (CASPAR). Some typical features of PsA are also observed in other chronic musculoskeletal diseases, as rheumatoid arthritis (RA) and HOA, determining possible delay of the diagnosis and consequent influence on the successful results of the therapies. In particular, the differential diagnosis of PsA and EHOA is very challenging, considering that both conditions can be characterized by bone proliferation and inflammation processes in the distal IP joints and lack of specific diagnostic biomarkers.

In the last decade, microRNA (miRNA) are emerged as possible candidate biomarkers in different rheumatic diseases. They are a class of small non-coding RNA molecules implicated in the direct regulation of the expression of different target genes by repressing or inhibiting translation. Mature miRNA are produced inside the cell and exert their function in the cytoplasm, but also by being released into the circulation and body fluids, where they regulate both physiological and pathological processes. Specific profiles of miRNA have been associated with the up-regulation of several inflammatory cytokines or degrading enzymes involved in the pathogenesis of PsA or OA. Indeed, miRNA have been detected in human plasma and in synovial fluid from patients with PsA and are considered possible diagnostic and prognostic biomarkers of this disease; very recently a pattern of circulating miRNAs has been studied also in patients with HOA.

IThe aim of the present study is to test whether miRNA can help to differentiate EHOA from PsA. In detail, the investigators evaluate the expression profile of a series of miRNA (miR-21, miR-140, miR-146a, miR-155, miR-181a, miR-223, miR-23a, miR-26a and miR-let-7e), known to be dysregulated in PsA and OA, in peripheral blood mononuclear cells (PBMCs) of patients with EHOA and PsA and in comparison to a group of healthy controls (HC).

Furthermore, the investigators assess the potential correlation between miRNA expression and disease activity.

ELIGIBILITY:
Inclusion Criteria:

For EHOA group:

* Diagnosis of EHOA according to the American College of Rheumatology (ACR) criteria and to the presence of the classical central erosion in at least two IP joints.
* Availability of plain radiography of both hands performed in the previous 6 months. Plain radiographs of both hands were collected and scored by two readers according to Kallman's classificationin a blind observation.

For PsA group:

* Diagnosis of PsA following the CASPAR classification guidelines
* peripheral arthritis pattern
* concomitant diagnosis of psoriasis confirmed by an expert dermatologist
* Naive to conventional and biologic disease-modifying anti-rheumatic drugs (DMARDs) or have withdrawn any DMARDs for at least three months, because of inadequate response or intolerance.

For control group:

* Healthy volunteers age-and sex-matched to study patients recruited among the hospital staff
* no symptoms or signs attributable to OA, psoriasis, as well as to autoimmune disorders and systemic inflammatory arthropathies.

Exclusion Criteria:

For all subjects:

* other rheumatic and not rheumatic diseases which can affect the functionality of the peripheral joints, as tendinopathies, carpal tunnel syndrome, Dupuytren's contractures, collagen diseases, neurological disorders or arthroplasty of the upper and lower limbs, recent trauma, or surgery of the concerned joints
* presence of inflammatory bowel diseases, liver or kidney diseases, acute or chronic infectious disorders, malignancy in the previous 5 years, pregnancy and breastfeeding.
* treatment with systemic or intra-articular (i.a.) corticosteroids, or with i.a. hyaluronic acid during the last three months.
* treatment with intra-muscular or intra-venous bisphosphonates in the previous 6 months

For EHOA group:

- therapy with Symptomatic Slow Acting Drugs for Osteoarthritis (SYSADOAs) during the previous 6 months.

For PsA group:

- PsA with pure axial involvement on the basis of inflammatory spinal pain and/or sacroiliac syndrome with spinal or sacroiliac radiographic changes and mixed involvement.

Ages: 40 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population included patients with erosive hand osteoarthritis, patients with psoriatic arthritis and healthy volunteers
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
MicroRNA expression profile | Baseline
  miR-21, miR-140, miR-146a, miR-155, miR-181a, miR-223, miR-23a, miR-26a and miR-let-7e expression in peripheral blood mononuclear cells

CONTACTS AND LOCATIONS:
Locations (1):
- Rheumatology Unit Azienda Ospedaliera Universitaria Senese, Siena, Italy

IPD SHARING:
Plan to Share IPD: No